CLINICAL TRIAL: NCT03737565
Title: Prospective, Multicenter and Observational Registry for the Evaluation of the Safety and Efficacy of Titanium-nitric Oxide-coated Stent (Optimax®) in Patients With Lesions With a Low Risk of Restenosis (Diameter ≥ 3.0 mm and Length ≤ 20 mm) (Reto 320 Study)
Brief Title: Evaluation of the Safety and Efficacy of Titanium-nitric Oxide-coated Stent (Optimax®) in Patients With Lesions With a Low Risk of Restenosis (Diameter ≥ 3.0 mm and Length ≤ 20 mm)
Acronym: RETO 320
Status: Completed | Type: Observational
Sponsor: Fundación EPIC (Other)
Responsible Party: Sponsor
Other Study IDs: RETO 320
Record Dates: First submitted 2018-11-08; First posted 2018-11-09 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-03

CONDITIONS: Coronary Artery Disease
Keywords: Cobalt-chromium
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Coronary Artery Disease
  Interventions: Device: Optimax stent®

INTERVENTIONS:
Device: Optimax stent® — Percutaneous coronary intervention with Optimax stent®

SUMMARY:
This prospective registry is intended to evaluate the safety and efficacy of the Optimax® stent.

DETAILED DESCRIPTION:
This prospective registry is intended to evaluate the safety and efficacy of the Optimax® stent in de novo coronary lesions with reference diameter ≥ 3.0 mm and Length ≤ 20 mm.

ELIGIBILITY:
Inclusion Criteria:

* Patients with age ≥ 18 years old.
* Patients with de novo coronary lesion treated with Optimax® stent, reference diameter = 3.0 mm and length ≤ 20 mm.
* Informed consent signed.

Exclusion Criteria:

* Refusal of the patient to participate at the study.
* Treatment of other injuries that do not meet the conditions (3x20).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with de novo coronary lesion treated with Optimax® stent, reference diameter = 3.0 mm and length ≤ 20 mm.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2019-02-17 (Actual); Primary Completion 2025-01-02 (Actual); Study Completion 2025-01-02 (Actual)

PRIMARY OUTCOMES:
Safety. The number of composite events of cardiac. | 6 and 12 month
  The number of composite events of cardiac death, myocardial infarction (MI) and stent thrombosis (Academic Research Consortium definitive/probable).
Efficacy: Incidence of clinically driven target lesion revascularization (TLR). | 6 and 12 month
  Incidence of clinically driven target lesion revascularization (TLR).Defined as any repeat percutaneous intervention of the target lesion or bypass surgery of the target vessel performed for restenosis or other complication of the target lesion.

SECONDARY OUTCOMES:
All death. | 6 and 12 month
  Systemic embolism, Major bleeding event (BARC ≥ 2).
Cardiac death. | 6 and 12 month
  Cardiac death.
Target Vessel revascularization. | 6 and 12 month
  Target Vessel revascularization.
Target lesion revascularization. | 6 and 12 month
  Target lesion revascularization.
Stent thrombosis (ARC definite/probable). | 6 and 12 month
  Stent thrombosis (ARC definite/probable).
Major bleeding event (BARC type 2-5). | 6 and 12 month
  Major bleeding event (BARC type 2-5).
Stroke. | 6 and 12 month
  Stroke.

CONTACTS AND LOCATIONS:
Locations (5):
- Spain (5):
  - Hospital de Mérida, Mérida, Badajoz
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital San Pedro de Alcántara, Cáceres
  - Hospital Universitario de León, León
  - Hospital Universitari Arnau de Vilanova, Lleida

REFERENCES:
- [Result] Lopez-Minguez JR, Nogales-Asensio JM, Romani S, Rivero-Crespo F, Aragon-Extremera VM, Jimenez-Mazuecos JM, Carrasco F, Oteo-Dominguez JF, Bosa-Ojeda F, Gomez-Hospital JA. TIOMAX: A Spanish Multicenter Registry of the real-world use of the TItanium OptiMAX(R) biostent: TIOMAX: Registro Espanol Multicentrico Del Biostent De Titanio OptiMAX(R) En La Vida Real. Catheter Cardiovasc Interv. 2018 Aug 1;92(2):261-268. doi: 10.1002/ccd.27326. Epub 2017 Sep 30. PMID 28963751
- [Result] Karjalainen PP, Nammas W, Ylitalo A, de Bruyne B, Lalmand J, de Belder A, Rivero-Crespo F, Kervinen K, Airaksinen JKE. Long-term clinical outcome of titanium-nitride-oxide-coated stents versus everolimus-eluting stents in acute coronary syndrome: Final report of the BASE ACS trial. Int J Cardiol. 2016 Nov 1;222:275-280. doi: 10.1016/j.ijcard.2016.07.267. Epub 2016 Aug 1. PMID 27497110
- [Result] Colkesen EB, Eefting FD, Rensing BJ, Suttorp MJ, Ten Berg JM, Karjalainen PP, Van Der Heyden JA. TIDES-ACS Trial: comparison of titanium-nitride-oxide coated bio-active-stent to the drug (everolimus)-eluting stent in acute coronary syndrome. Study design and objectives. Minerva Cardioangiol. 2015 Feb;63(1):21-9. PMID 25670057